CLINICAL TRIAL: NCT01417533
Title: A Natural History Study of Patients With GNE Myopathy and GNE-Related Diseases
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Collaborators: Therapeutics for Rare and Neglected Diseases (TRND) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110218; 11-HG-0218
Record Dates: First submitted 2011-08-13; First posted 2011-08-16 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11-19

CONDITIONS: GNE Myopathy; GNE Related Diseases
Keywords: Hereditary Inclusion Body Myopathy; Natural History
MeSH Terms: conditions — Distal myopathy, Nonaka type

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GNE: Patients with a diagnosis of GNE myopathy
- GNE-Related Diseases: Patient with a GNE related disease
- non-GNE: Subjects that are a carrier family member or a caregiver of a patient on the study are eligibleto participate.

SUMMARY:
Background:

- GNE Myopathy is a disease that causes walking difficulties and increasing muscle weakness. It usually develops in young adults (between 20 and 30 years of age), and affects arm and leg muscles. HIBM is caused by mutations in a gene that may affect how the muscles function. Researchers want to learn more about the causes, symptoms, and effects of HIBM.

Objectives:

- To collect genetic and medical information from people with GNE Myopathy .

Eligibility:

- Individuals between 18 and 80 years of age who have GNE Myopathy and do not use a wheelchair. - Participants must be willing to stop any current treatment of HIBM while enrolled in the study.

Design:

* Participants will be screened with a medical history, physical exam, and neurological exam.
* At the first visit, participants will have the following tests:
* Questionnaires about the impact of HIBM on daily activities, mood, and quality of life
* 24-hour urine collection
* Blood samples
* Heart function tests
* Muscle strength and endurance tests, including walking
* Imaging study of the muscles
* Participants will return for followup visits at 6, 12, and 18 months. They may be asked to return for a final visit at 24 months. Not all tests will be performed at each visit.
* Treatment will not be provided as part of this protocol.

For more information, visit our website: http://hibmstudy.nhgri.nih.gov/

DETAILED DESCRIPTION:
This is a prospective observational study to evaluate patients with GNE myopathy and other GNE-related diseases. The GNE gene encodes for UDP-GlcNAc 2-epimerase/ManNAc kinase, the bifunctional enzyme that initiates and regulates intracellular sialic acid (Neu5Ac) biosynthesis and glycan sialylation. GNE myopathy is a rare, autosomal recessive myopathy with onset in early adulthood characterized by progressive skeletal muscle atrophy and weakness. The impairment of Neu5Ac production is presumed to cause decreased sialylation of muscle glycoproteins, resulting in muscle deterioration. Other GNE-related diseases such as congenital thrombocytopenia have been recently identified, but the pathophysiology is not well understood. In this protocol, we plan to evaluate patients with GNE myopathy and other GNE-related diseases clinically, biochemically, and molecularly to characterize the mechanisms of disease, to delineate the natural history, phenotypes, progression and complications of GNE-related diseases, and to identify endpoints and biomarkers to support clinical trials testing potential therapies.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 4-80 years, either gender, inclusive.
  2. Diagnosis of GNE myopathy or GNE-related diseases based upon the identification of GNE gene mutations. Molecular confirmation of the diagnosis will be obtained for all subjects in the study.
  3. Subjects that are a carrier family member of a patient on the study are eligible to participate.
  4. Must be able to provide informed consent.

EXCLUSION CRITERIA:

1. Psychiatric illness or other diseases that would interfere with the subject s ability to comply with the requirements of this protocol.
2. Hepatic laboratory parameters (aspartate aminotransferase [AST], alanine aminotransferase [ALT]) or renal laboratory parameters (creatinine, blood urea nitrogen [BUN]) greater than 3 times the upper limit of normal.
3. Presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, metabolic, or gastrointestinal disease not related to the primary disease process.

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of GNE myopathy or GNE-related disease. Subjects that are a carrier family member or a caregiver of a patient on the study are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2011-09-14 (Actual)

PRIMARY OUTCOMES:
Natural History | Ongiong
  To delineate the natural history of GNE myopathy, and to further characterize the phenotype, progression and complications of the disease.

SECONDARY OUTCOMES:
Endpoints | Ongoing
  To identify endpoints and biomarkers of the disease. To study factors that contribute to disease heterogeneity.

CONTACTS AND LOCATIONS:
Overall Officials: William A Gahl, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Liu CY, Yao J, Kovacs WC, Shrader JA, Joe G, Ouwerkerk R, Mankodi AK, Gahl WA, Summers RM, Carrillo N. Skeletal Muscle Magnetic Resonance Biomarkers in GNE Myopathy. Neurology. 2021 Feb 2;96(5):e798-e808. doi: 10.1212/WNL.0000000000011231. Epub 2020 Nov 20. PMID 33219145
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-HG-0218.html